CLINICAL TRIAL: NCT04237636
Title: A Clinical Score to Predict Acute Kidney Injury After Heart Valve Replacement
Brief Title: A Clinical Score to Predict Acute Kidney Injury After Heart Valve Replacement Surgery
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, chonglei, MD& PhD, Xijing Hospital
Other Study IDs: KY20192157-C-1
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with post-operative AKI: Patients developing acute kidney injury (AKI) following heart valve replacement surgery.
  AKI was classified according to the KDIGO definition[10]. Stage-1 AKI: increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.5μmol/l) or increase to more than or equal to 150% to 200% (1.5≤x<2) from baseline within 7 days. Stage-2 AKI: Increase in serum creatinine to more than 200% to 300% (2≤x<3) from baseline. Stage-3 AKI: Increase in serum creatinine to more than 300% (3≤) from baseline (or serum creatinine of more than or equal to 4.0 mg/dl (≥ 353.6μmol/l) or when the patient commenced RRT.
- Patients without post-operative AKI: Patients with normal kidney function (without acute kidney injury (AKI)) following heart valve replacement surgery

SUMMARY:
Acute kidney injury (AKI) is a common and severe complication of cardiac surgery. The main stay treatment remains preventive with no clear evidence supporting any therapeutic interventions. AKI risk prediction scores are an objective, transparent means of cohort enrichment but are not widely used. The purpose of this analysis was to develop and validate a clinical score including pre-,intra-and post-operative predictors that predicted AKI following heart valve replacement surgery. This prediction score allows identification of patients at high risk of AKI and may support decision-making for protective kidney treatment.

DETAILED DESCRIPTION:
This study is a single center retrospective observational study designed to to develop and validate a clinical score that predicts AKI after heart valve replacement surgery。 To achieve this goal, patient underwent heart valve replacement surgery will be screened for enrollment eligibility. For the purpose of this analysis, only the first surgical episode was considered. Patients required preoperative dialysis, with any degree of renal insufficiency (acute or chronic) and patients who had end-stage renal disease (estimated glomerular fltration rate [eGFR] < 15 mL/min /1.73m2 )are not included in study.

AKI was classified according to the KDIGO definition[10]. Stage-1 AKI: increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.5μmol/l) or increase to more than or equal to 150% to 200% (1.5≤x<2) from baseline within 7 days. Stage-2 AKI: Increase in serum creatinine to more than 200% to 300% (2≤x<3) from baseline. Stage-3 AKI: Increase in serum creatinine to more than 300% (3≤) from baseline (or serum creatinine of more than or equal to 4.0 mg/dl (≥ 353.6μmol/l) or when the patient commenced RRT.

We selected demographic, preoperative, intra-operative and early postoperative variables considered predictors of AKI.

1. The demographic and preoperative factors included age, sex, weight, height; history of smoke, drink, angina, cerebrovascular disease, COPD, peripheral vascular disease, hypertension, valve infection , arrythmia , diabetes mellitus, MI , atrial fibrillation, pulmonary hypertension, previous cardiac surgery; NYHA stage, surgery type , Operative approach and emergency surgery。The latest value before operation: serum creatinine level, haemoglobin, capillary glucose, hemoglobin，WBC, EF, LDL-C , urinary protein, CRP, PCT, ALB, TBIL, PT and Glomerular filtration rate (GFR). History of taking the following drugs before surgery: contrast, nephrotoxic antibiotics, β-blocker, calcium channel blocker, lasix, ACEI, ARB, immunosuppressive, heparin, aspirin, clopidogrel, ticagrelor, digoxin, levosimendan, dopamine, dobutamine, cedilanid, isosorbide dinitrate, isosorbide mononitrate, isoprenaline and NASID.
2. The intra-operative factors included cardiopulmonary bypass time, cross-clamp time, transfusion, FFP, VFP, CFP，output and input ; the highest blood glucose, minimum hematocrit, minimum mean arterial pressure, minimum temperature and fluid balance during CPB.
3. The postoperative factors included time to extubation, mean ICU and hospital stay and mortality. First measured value after entering ICU: CVP, PH, HB.

We also considered postoperative complications during the intensive care unit included IABP, ECMO, cardiac arrest, arrhythmia, re-intubation, return to ICU，tracheotomy.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Subjects undergoing heart valve replacement surgery

Exclusion Criteria:

* Pregnancy
* Transplant donor or recipient
* Required preoperative dialysis, with any degree of renal insufficiency (acute or chronic) and patients who had end-stage renal disease (estimated glomerular fltration rate [eGFR] < 15 mL/min /1.73m2 )
* Local anesthesia
* Lack of creatinine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We included adult patients undergoing heart valve replacement surgery between January first, 2014 and December 31, 2018 in a single tertiary hospital (Xijing Hospital, Xi'an, China)
Sampling Method: Non-Probability Sample
Enrollment: 3392 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Development of an prediction score for AKI(including stage 1,2 and 3) | during postoperative day 7
  Development of an simple and easy applicable score based on pre-，intra-and post-operative risk factors to predict postoperative AKI in patients for heart valve replacement surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, MD, PhD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Zacharias M, Gilmore IC, Herbison GP, Sivalingam P, Walker RJ. Interventions for protecting renal function in the perioperative period. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD003590. doi: 10.1002/14651858.CD003590.pub2. PMID 16034904
- [Background] Birnie K, Verheyden V, Pagano D, Bhabra M, Tilling K, Sterne JA, Murphy GJ; UK AKI in Cardiac Surgery Collaborators. Predictive models for kidney disease: improving global outcomes (KDIGO) defined acute kidney injury in UK cardiac surgery. Crit Care. 2014 Nov 20;18(6):606. doi: 10.1186/s13054-014-0606-x. PMID 25673427
- [Background] Thakar CV, Arrigain S, Worley S, Yared JP, Paganini EP. A clinical score to predict acute renal failure after cardiac surgery. J Am Soc Nephrol. 2005 Jan;16(1):162-8. doi: 10.1681/ASN.2004040331. Epub 2004 Nov 24. PMID 15563569
- [Background] Mehta RH, Grab JD, O'Brien SM, Bridges CR, Gammie JS, Haan CK, Ferguson TB, Peterson ED; Society of Thoracic Surgeons National Cardiac Surgery Database Investigators. Bedside tool for predicting the risk of postoperative dialysis in patients undergoing cardiac surgery. Circulation. 2006 Nov 21;114(21):2208-16; quiz 2208. doi: 10.1161/CIRCULATIONAHA.106.635573. Epub 2006 Nov 6. PMID 17088458
- [Background] Huen SC, Parikh CR. Predicting acute kidney injury after cardiac surgery: a systematic review. Ann Thorac Surg. 2012 Jan;93(1):337-47. doi: 10.1016/j.athoracsur.2011.09.010. PMID 22186469
- [Background] Lassnigg A, Schmidlin D, Mouhieddine M, Bachmann LM, Druml W, Bauer P, Hiesmayr M. Minimal changes of serum creatinine predict prognosis in patients after cardiothoracic surgery: a prospective cohort study. J Am Soc Nephrol. 2004 Jun;15(6):1597-605. doi: 10.1097/01.asn.0000130340.93930.dd. PMID 15153571
- [Background] Jorge-Monjas P, Bustamante-Munguira J, Lorenzo M, Heredia-Rodriguez M, Fierro I, Gomez-Sanchez E, Hernandez A, Alvarez FJ, Bermejo-Martin JF, Gomez-Pesquera E, Gomez-Herreras JI, Tamayo E. Predicting cardiac surgery-associated acute kidney injury: The CRATE score. J Crit Care. 2016 Feb;31(1):130-8. doi: 10.1016/j.jcrc.2015.11.004. Epub 2015 Nov 6. PMID 26700607
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Brown JR, Cochran RP, Leavitt BJ, Dacey LJ, Ross CS, MacKenzie TA, Kunzelman KS, Kramer RS, Hernandez F Jr, Helm RE, Westbrook BM, Dunton RF, Malenka DJ, O'Connor GT; Northern New England Cardiovascular Disease Study Group. Multivariable prediction of renal insufficiency developing after cardiac surgery. Circulation. 2007 Sep 11;116(11 Suppl):I139-43. doi: 10.1161/CIRCULATIONAHA.106.677070. PMID 17846294
- [Derived] Yan Y, Gong H, Hu J, Wu D, Zheng Z, Wang L, Lei C. Perioperative parameters-based prediction model for acute kidney injury in Chinese population following valvular surgery. Front Cardiovasc Med. 2023 Mar 7;10:1094997. doi: 10.3389/fcvm.2023.1094997. eCollection 2023. PMID 36960471